CLINICAL TRIAL: NCT00062686
Title: An Open-Label, Multicenter, Single Arm Phase II Study of Oral GW572016 as Single Agent Therapy in Subjects With Advanced or Metastatic Breast Cancer Who Have Progressed While Receiving HERCEPTIN-Containing Regimens
Brief Title: GW572016 For Treatment Of Refractory Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EGF20008; NCT00068627 (obsolete NCT alias)
Record Dates: First submitted 2003-06-11; First posted 2003-06-12 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Neoplasms, Breast
Keywords: Lapatinib; Metastatic Breast Cancer; HERCEPTIN refractory
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GW572016

SUMMARY:
This study was designed to determine the efficacy of an oral dual kinase inhibitor for the treatment of metastatic breast cancer tumors that are known to overexpress ErbB2 in a refractory patient population.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent.
* Histologically confirmed Stage IIIb or IV breast cancer.
* Refractory breast cancer defined as progression in the metastatic setting after prior therapy with anthracyclines, taxanes and capecitibine.
* Subjects with documented ErbB2 tumor overexpression must have received at least 6 cycles of trastuzumab.
* Documented disease progression of the most recent treatment is required.
* Archived tumor tissue available for testing.
* Measurable lesions according to Response Evaluation Criteria In Solid Tumors (RECIST).
* At least 3 weeks since prior cancer therapies except for trastuzumab which must be discontinued at least 2 weeks prior to the beginning of study drug.
* Bisphosphonate therapy initiated prior to study entry is allowed, however, initiation of bisphosphonates following study entry is not allowed.
* Able to swallow and retain oral medication.
* Cardiac ejection fraction within the institutional normal range as measured by echocardiogram or MUGA (Multiple Gated Acquisition) scan.
* Adequate kidney and liver function.
* Adequate bone marrow function.

Exclusion criteria:

* Pregnant or lactating.
* Copies of nadir scans and/or photographs of the tumor prior to disease progression as well as scans documenting disease progression are not available for review.
* Malabsorption syndrome, ulcerative colitis, disease significantly affecting gastrointestinal function or resection of the stomach or small bowel.
* History of other malignancy.
* Serious medical or psychiatric disorder that would interfere with the patient''s safety or informed consent.
* Active or uncontrolled infection.
* Known history of uncontrolled or symptomatic angina, arrhythmias or congestive heart failure.
* Known history of or clinical evidence of leptomeningeal carcinomatosis.
* Active infection.
* Concurrent cancer therapy or investigational therapy.
* Use of oral or IV steroids.
* Unresolved or unstable serious toxicity from prior therapy.
* Prior treatment with an ErbB1 and/or ERbB2 inhibitor other than trastuzumab.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2003-11; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Tumor response rate

SECONDARY OUTCOMES:
clinical benefit rate time to progression 4 and 6 month progression free survival overall survival

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- GSK Investigational Site, Buenos Aires, Buenos Aires, Argentina
- GSK Investigational Site, Villejuif, France
- GSK Investigational Site, Augsburg, Bavaria, Germany
- United Kingdom (4):
  - GSK Investigational Site, Sutton, Surrey
  - GSK Investigational Site, Bebington, Wirral
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester